CLINICAL TRIAL: NCT02705365
Title: Patient Navigation for Lung Screening at MGH Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sanja Percac-Lima, MD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015P002239; CCCDAA-14-012-01-CCCDA (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Lung Cancer
Keywords: Lung Screening; Low-Dose Computer Tomography; Patient Navigation
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigation (Experimental): Patients assigned to the patient navigator (PN) arm will be sent a letter about the program with lung screening educational materials. The PN will educate eligible patients about lung screening, explore barriers to screening, coordinate scheduling an appointment with a provider, and possibly attend the visit with the patient. The PN will further coordinate scheduling the CT scan, help the patient obtain the test, and access any required follow-up. The PN will assess the patient's interest in quitting smoking and if so, offer and help to connect the smoker to existing cessation resources in the community and provide follow-up contacts to monitor adherence to treatments.
  Interventions: Other: Patient Navigation
- Usual Care (Active Comparator): The control group will receive usual care during the 1-year study period. After the study period, they will be offered 1:1 patient navigation to obtain lung screening and follow-up of abnormal results as well as smoking cessation guidance.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Patient Navigation — One to one patient navigation to obtain lung screening and follow-up of abnormal results, as well as smoking cessation guidance.
  Arms: Patient Navigation
Other: Usual Care — Usual care during the study period. After the study period, they will be offered 1:1 patient navigation to obtain lung screening and follow-up of abnormal results, as well as smoking cessation guidance.
  Arms: Usual Care

SUMMARY:
To develop and implement a patient navigator (PN) program for lung screening and smoking cessation in community health center primary care practices. This program will be evaluated in a randomized controlled trial of primary care patients who currently smoke.

DETAILED DESCRIPTION:
The specific aims of this study are:

Specific Aim 1: To develop a patient navigator (PN) program for lung screening for patients who are current smokers, aged 55-77 years, potentially eligible for lung screening and are receiving care at community health centers (CHCs) affiliated with MGH.

Specific Aim 2: To evaluate the effectiveness of the new lung screening PN program in improving screening rates and increasing use of tobacco cessation services in a randomized controlled trial.

Specific Aim 3: To demonstrate that equity is maintained in rates of lung screening and in follow up of abnormal chest CT results, comparing eligible smokers from CHCs with eligible smokers from other practices within the MGH primary care network.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients aged 55-77 years who are current cigarette smokers (according to an algorithm using electronic medical record data), and
2. receive care at one of the five Massachusetts General Hospital community health centers.

Exclusion Criteria:

1. patients who have previously received a diagnosis of lung cancer,
2. have undergone a chest CT within 18 months before enrollment,
3. are subsequently identified as having died prior to the study intervention,
4. deemed by their primary care provider as not eligible for lung screening.

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Percac-Lima, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Percac-Lima S, Ashburner JM, Rigotti NA, Park ER, Chang Y, Kuchukhidze S, Atlas SJ. Patient navigation for lung cancer screening among current smokers in community health centers a randomized controlled trial. Cancer Med. 2018 Mar;7(3):894-902. doi: 10.1002/cam4.1297. Epub 2018 Feb 21. PMID 29464877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Navigation | Usual Care
Started | 400 | 800
Completed | 400 | 800
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigation | Usual Care | Total
Number analyzed (Participants) | 400 | 800 | 1200
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (5.4) | 62.4 (5.7) | 62.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 442 | 630
  Male | 212 | 358 | 570
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 22 | 40
  Black | 18 | 25 | 43
  Hispanic | 26 | 41 | 67
  Other/Unknown | 27 | 46 | 73
  White | 311 | 666 | 977
Language [Count of Participants; unit: Participants]
  English | 352 | 714 | 1066
  Non-English | 48 | 86 | 134
Insurance [Count of Participants; unit: Participants]
  Commercial | 128 | 280 | 408
  Medicare | 47 | 84 | 131
  Medicaid | 121 | 211 | 332
  Dual Medicare/Medicaid | 103 | 225 | 328
  Self | 1 | 0 | 1
Clinic Visits Over 3 Years [Mean (Standard Deviation); unit: visits] | 10.3 (7.9) | 10.7 (8.4) | 10.5 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Chest CT Completion
Description: Percentage of patients assigned to the intervention and control groups who had at least one chest CT (according to billing and EMR data) during the 1-year study period.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation | Usual Care
Number analyzed (Participants) | 400 | 800
Participants | 124 | 138

2. Secondary Outcome: Tobacco Treatment Use
Description: Percentage of patients, comparing intervention and control groups, who during the 1-year study period had referral to Massachusetts Quitline, smoking cessation medication prescribed, or referral to in-person counseling.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation | Usual Care
Number analyzed (Participants) | 400 | 800
Participants | 133 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Patient Navigation | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/800
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/800
Other Adverse Events (participants affected / at risk) | 0/400 | 0/800

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT02705365/Prot_SAP_000.pdf